CLINICAL TRIAL: NCT05926674
Title: Immediate Effects of Myofascial Release on Lumbar Range of Motion. A Randomized Control Trial.
Brief Title: Does Manual Therapy Provide Immediate Improvement in Lumbar Range of Motion?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York Institute of Technology (Other)
Responsible Party: Principal Investigator, Mark Gugliotti, Doctor, New York Institute of Technology
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BHS-1851
Record Dates: First submitted 2023-06-07; First posted 2023-07-03 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: N/A Healthy Individuals
MeSH Terms: interventions — Myofascial Release Therapy

STUDY DESIGN:
Intervention Model Description: This study is a double-arm repeated measures study performed in a single session lasting approximately 30-40 minutes.
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessors will not have knowledge of each participant's intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Myofascial Release (Experimental): Myofascial release (MFR) is a manual therapy technique commonly used by clinicians and bodyworkers to provide effects such as decreased pain, improvement in flexibility, ROM, and quality of life. It combines non-gliding fascial traction with varying amounts of stretching to produce a tensional force on the muscle and its associated fascia resulting in viscoelastic lengthening and deformation.
  Myofascial release will be provided to each subject assigned to the experimental group by the primary investigator (PI). The participant will be positioned in prone and the MFR will be applied along the lumbar paraspinals bilaterally for five minutes per side.
  Interventions: Other: Myofascial Release
- Light Touch Contact (Sham Comparator): Sham treatment will be provided to each subject assigned to the control group by the designated co-investigator. The sham treatment of light touch will be applied to the lumbar paraspinals in the same fashion as noted above. This form of light touch contact is not therapeutic and is meant to only mimic a manual therapy technique.
  Interventions: Other: Light Touch Contact

INTERVENTIONS:
Other: Myofascial Release — Myofascial release is a manual therapy technique commonly used by clinicians and bodyworkers to provide effects such as decreased pain, improvement in flexibility, ROM, and quality of life. It combines non-gliding fascial traction with varying amounts of stretching to produce a tensional force on the muscle and its associated fascia resulting in viscoelastic lengthening and deformation.
  Arms: Myofascial Release
Other: Light Touch Contact — The sham treatment of light touch will be applied to the lumbar spine and this form of contact is not therapeutic. It is only meant to only mimic a manual therapy technique.
  Arms: Light Touch Contact

SUMMARY:
The goal of this clinical study is to determine if manual therapy can improve lumbar mobility in healthy individuals.

The main questions it aims to answer are:

* Is there an immediate local spinal effect?
* Is there an associated distal effect?

Researchers will compare an experimental group and a control group to examine the effects.

DETAILED DESCRIPTION:
Upon consent, participants will be assessed for lumbar spine mobility using inclinometers, hamstring flexibility using the active knee extension test and the modified sit-and-reach test, and ease of lifting a small, weighted object. After baseline measures are recorded, the participants will receive an intervention that will be either therapeutic (myofascial release) or sham (non-therapeutic hand placement). The choice of intervention received will be previously determined through the use of randomization software. The intervention provided will be applied to the low back and last for a total of 10 minutes. Immediately following the intervention, participants will again be assessed for lumbar spine mobility, hamstring flexibility, and ease of lifting a small, weighted object as noted above.

ELIGIBILITY:
Inclusion Criteria:

* New York Institute of Technology students
* At least 18 years old
* Good overall health

Exclusion Criteria:

* Pacemaker
* Any previous history of lumbar or connective tissue pathology
* Down syndrome
* Prolonged steroid use
* Oswestry Low Back Disability score of >10 (ODI)
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-07-26 (Actual)

PRIMARY OUTCOMES:
Lumbar Range of Motion | 3 minutes
  Upon arrival, the participant will be greeted and directed to the research room. The participant will be instructed to stand comfortably with their feet shoulder width apart, followed by one inclinometer placed at the level of S2 and the other 15cm above S2 by the designated researcher. The placement of the inclinometers is necessary to establish proper measurement of the lumbar spine, independent of outside influence. Inclinometers are valid and reliable tools for measuring lumbar ROM. Lumbar flexion will be measured first, followed by lateral flexion to the left and right. Lumbar ROM will be measured before and after each treatment.
Modified Sit and Reach test | 3 minutes
  The modified sit and reach test is a valid and reliable tool for assessing hamstring flexibility. This assessment will be implemented by the designated researcher. The modified sit and reach test will be administered before and after each treatment.
Active Knee Extension test | 3 minutes
  The test is performed supine with the tested leg bent to 90° of supported hip flexion. The participant will be asked to actively extend his or her knee as fully as possible. Any lag from full extension will be measured with a standard goniometer. This test is a valid and reliable tool for hamstring length assessment. An extension lag of greater than 20° indicates a lack of hamstring flexibility. This will be performed on both lower extremities before and after each treatment.
Functional Movement Assessment | 1 minute
  Each participant will be asked to perform a low-level functional activity (picking up a light-weight object) to help identify any perceived change in ability following the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Gugliotti, DPT, Principal Investigator — New York Institute of Technology
Locations (1):
- NYIT, Old Westbury, New York, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD for this study.